CLINICAL TRIAL: NCT04449003
Title: Influence of Stress and Psychiatric Symptoms on Children With Tourette Syndrome
Acronym: InSPSCTS
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Isaacs, Assistant Professor of Neurology, Vanderbilt University Medical Center
Other Study IDs: U11234
Record Dates: First submitted 2020-06-20; First posted 2020-06-26 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Tourette Syndrome in Adolescence; Tourette Syndrome; Tourette Syndrome in Children
Keywords: Stress; Self-esteem; Quality of life
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents with Tourette Syndrome: Adolescents (aged 13-17 years) with Tourette Syndrome
- Adolescents without any neurologic or psychiatric diagnoses: Adolescents (aged 13-17 years) without any history of tics

SUMMARY:
Investigators propose a cross-sectional, observational pilot study to examine the contribution of stress, family dynamics, and peer relationships to quality of life (QOL) in adolescents with Tourette syndrome (TS). Investigators will recruit two groups of participants: 1) adolescents aged 13-17 years of age with TS and 2) adolescents aged 13-17 without any neurologic or psychiatric diagnoses. Participants and one of their parents/caregivers will complete a series of questionnaires screening for and quantifying the extent of stress and mental health symptoms, including anxiety, depression, obsessive compulsive disorder (OCD), attention deficit hyperactivity disorder (ADHD). Participants will also complete instruments characterizing family interactions and peer relationships. Adolescents with TS will also undergo a semi-structured interview assessing the severity of their tics.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a multi-faceted neurodevelopmental disorder with wide-ranging impact on adolescent quality of life (QOL). Comorbid psychiatric and psychological factors exert greater influence on QOL than tics in TS, but the specific role of stress, family dynamics, and peer relationships has been largely overlooked, despite the fact that these factors are known to impact QOL in those with chronic disease. Investigators propose a cross-sectional, observational pilot study to examine the contribution of stress, family dynamics, and peer relationships to QOL in adolescents with TS. The primary goal of this study is to collect sufficient data for hypothesis-generation and power analysis refinement in planning of a larger scale study.

Investigators will recruit adolescents aged 13-17 years of age with TS presenting for regular care at the Vanderbilt Pediatric Neurology Clinic. Adolescents without any neurologic or psychiatric diagnoses will be recruited as a control population. Participants and one of their parents/caregivers will complete a series of questionnaires screening for and quantifying the extent of stress and mental health symptoms, including anxiety, depression, obsessive compulsive disorder (OCD), attention deficit hyperactivity disorder (ADHD). Participants will also complete instruments characterizing family interactions and peer relationships. The scale battery can be completed by the adolescent and caregiver in parallel and is anticipated to take 60-75 minutes total to complete. Adolescents with TS will also undergo a semi-structured interview assessing the severity of their tics. The study plans to enroll subjects over a 12-month time frame.

ELIGIBILITY:
Inclusion Criteria for adolescents with TS:

* adolescent age 13-17 years of age
* adolescent diagnosis of Tourette syndrome (TS)
* English-speaking adolescent and caregiver (as validated questionnaires are in English)
* adolescent and caregiver willingness and ability to complete relevant questionnaires

Exclusion Criteria for adolescents with TS:

* cognitive or attentional impairment precluding ability of adolescent or caregiver to complete self-report questionnaires
* adolescent diagnosis of genetic conditions besides TS and its known comorbidities
* adolescent with severe medical conditions unrelated to TS (e.g. uncontrolled seizures, prominent heart conditions)

Inclusion Criteria for adolescents without any neurologic or psychiatric diagnoses:

* adolescent age 13-17 years of age
* no history of tics
* English-speaking adolescent and caregiver
* adolescent and caregiver willingness and ability to complete relevant questionnaires

Exclusion Criteria for adolescents without any neurologic or psychiatric diagnoses:

* cognitive or attentional impairment precluding ability of adolescent or caregiver to complete self-report questionnaires
* adolescent with severe medical conditions

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patient study population consists of adolescents aged 13-17 years of age with Tourette syndrome presenting for routine clinical care, as well as the adolescents' caregivers. The control study population consists of adolescents aged 13-17 years of age without tics, as well as the adolescents' caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Youth Quality of Life Research Version (YQOL-R) | Baseline
  Self-report quality of life scale comprised of 42 items with 10-point Likert scale (raw total score 0-420) and 15 additional items with open-ended and demographic questions. Higher scores indicate better overall quality of life.

SECONDARY OUTCOMES:
Cohen's Perceived Stress Scale | Baseline
  Self-report stress scale comprised of 10 items (total score range 0-40). Higher scores indicate greater perceived stress.
PedsQL - Family Impact Module | Baseline
  Caregiver-report scale comprised of 36 items (total score range 0-100) assessing impact of health condition(s) on family. Higher scores indicate better family functioning in context of health-related condition(s).
Conners-3 Parent Short QuikScore Forms | Baseline
  Caregiver-report scale comprised of 45 items assessing inattention, hyperactivity, and executive functioning of child. T-scores are generated, with higher scores indicating greater deviation from norms.
Revised Children's Anxiety and Depression Scale (RCADS) - Parent Report | Baseline
  Caregiver-report scale comprised of 47 items assessing mood symptoms. T-scores are generated, with higher scores indicating greater deviation from norms.
Revised Children's Anxiety and Depression Scale (RCADS) - Self-Report | Baseline
  Self-report scale comprised of 47 items assessing mood symptoms. T-scores are generated, with higher scores indicating greater deviation from norms.
Yale Global Tic Severity Scale (YGTSS) | Baseline
  Semi-structured clinician-administered interview assessing tic severity, with total tic score range of 0-50 and functional impairment scale range of 0-50. Higher scores indicate greater tic severity and functional impairment, respectively. This measure will only be administered to adolescents with TS.
School and Mental Health Services Inventory | Baseline
  Questionnaire assessing educational and functional status of child. No total score generated.
Rosenberg Self Esteem Scale | Baseline
  Self-report self-esteem scale comprised of 10 items (total score range 10-40). Higher scores indicate higher self-esteem.
Kearney's Daily Life Stressors Scale | Baseline
  Self-report scale consisting of 30 items (total score range 0-120) assessing degree of stress caused by daily activities. Higher scores indicate greater burden from daily stressors.
McMaster Family Assessment Device | Baseline
  Self-report scale consisting of 60 items (total score range 0-180) assessing structural, organizational, and interactional aspects of family environment. The scale contains subscales, the scores of which are added to create a composite overall score, with higher scores indicative of more supportive family environment.
PROMIS Peer Relationships Short Form 8a - Self Report | Baseline
  Self-report scale consisting of 8 items (total score is composite of individual item scores, ranked on Likert scale from 1-5) assessing quality of peer relationships. Total raw scores are converted to a T-score. Higher scores indicate more positive perception of peer relationships.
PROMIS Peer Relationships Short Form 8a - Proxy-Report | Baseline
  Proxy-report scale consisting of 8 items (total score is composite of individual item scores, ranked on Likert scale from 1-5) assessing quality of child's peer relationships. Total raw scores are converted to a T-score. Higher scores indicate more positive perception of child peer relationships.

CONTACTS AND LOCATIONS:
Overall Officials: David A Isaacs, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Heather Riordan, MD, Principal Investigator — Vanderbilt Children's Hospital
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided